CLINICAL TRIAL: NCT00233883
Title: An Open-label Study of the Tolerability of a Subcutaneous Needle-free Injection Device Used to Administer Fuzeon, Compared With the Standard Needle/Syringe Supplied With Commercial Fuzeon in HIV-1 Infected, ARV Treatment-experienced Adults
Brief Title: WAND Study - A Study to Evaluate Fuzeon (Enfuvirtide) Administered by a Needle-Free Injection Device in Patients With HIV.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Trimeris (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ML18596
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Enfuvirtide

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: enfuvirtide [Fuzeon]
- 2 (Active Comparator)
  Interventions: Drug: enfuvirtide [Fuzeon]

INTERVENTIONS:
Drug: enfuvirtide [Fuzeon] — 90mg sc bid by Biojector 2000 NFID for 4 weeks
  Arms: 1
Drug: enfuvirtide [Fuzeon] — 90mg sc bid by 27G1/2" needle/syringe for 4 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the tolerability of a subcutaneous needle-free injection device used to administer Fuzeon, compared with the standard needle/syringe supplied with commercial Fuzeon. The anticipated time on study treatment is <3 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients, >=18 years of age with HIV-1 infection;
* previously treated with antiretroviral agents.

Exclusion Criteria:

* prior use of Fuzeon or T-1249;
* inability to self-inject;
* active, untreated opportunistic infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2005-08; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Composite endpoint (pain, induration, nodules/cysts). | Throughout study

SECONDARY OUTCOMES:
Steady state C trough | Weekly
Signs and symptoms associated with Fuzeon injections | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- United States (14):
  - Long Beach, California
  - Los Angeles, California
  - Washington D.C., District of Columbia
  - Fort Lauderdale, Florida
  - South Miami, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Boston, Massachusetts
  - Detroit, Michigan
  - St Louis, Missouri
  - Winston-Salem, North Carolina
  - Dallas, Texas
  - Houston, Texas
  - Annandale, Virginia

REFERENCES:
- [Derived] Gottlieb M, Thommes JA; WAND Study Team. Short communication safety, tolerability and pharmacokinetics of enfuvirtide administered by a needle-free injection system compared with subcutaneous injection. Antivir Ther. 2008;13(5):723-7. PMID 18771056